CLINICAL TRIAL: NCT00936312
Title: Females With Severe or Moderate Hemophilia A or B: an International Multi-center Study
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Bayer (Industry); University Hospital, Bonn (Other)
Responsible Party: Sponsor
Other Study IDs: Intl Female Hemophilia Study
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Hemophilia A; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Females with Hemophilia: Females with severe or moderate Hemophilia A or B
- Control group: Male subjects with severe Hemophilia A or B and female subjects with mild (20-60%) Hemophilia A or B.

SUMMARY:
This is a multi-center, international study designed to collect clinical, genetic and quality of life information on females with hemophilia, an inherited bleeding disorder. The study is designed to determine whether there are problems and issues unique to females with hemophilia.

DETAILED DESCRIPTION:
The study involves two questionnaires: one on the diagnosis, symptoms, complications and treatment of each participant to be completed by a staff member; the other is a questionnaire to be completed by the participant on how the disease has affected her life. Finally, for those participants who have not previously had genetic testing, the third part of the study is an optional blood test to determine the genetic cause, what change in the factor VIII or factor IX gene, caused the hemophilia. The test results will be available to those participants who wish to learn their results. With the data we collect we will compile a database to examine the connection between the genetic cause of hemophilia and the course and symptoms of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Females with severe (FVIII<0.01u/ml) or moderate (FVIII 0.01≤0.05 u/ml) hemophilia A
* Females with severe (FIX<0.01u/ml) or moderate (FIX 0.01≤0.05u/ml) hemophilia B
* Willingness to participate in the study.

Exclusion Criteria:

* Subjects who do not meet the inclusion criteria with respect to gender or hemophilia severity.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Females with severe or moderate Hemophilia A (less than or equal to 5%) Females with severe or moderate Hemophilia B (less than or equal to 5%)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The molecular and cytogenetic etiology of the condition will be compiled. Clinical manifestation demonstrated by the female hemophiliacs will be compared to published data available. Genotype and phenotype will be correlated. | 1-2 visits

CONTACTS AND LOCATIONS:
Overall Officials: William B Mitchell, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (11):
- Weill Cornell Medical College, New York, New York, United States
- Princess Margaret Hospital for Children, Perth, Australia
- Germany (2):
  - University Clinic Bonn, Bonn
  - University Clinic Munich, Munich
- Sheba Medical Center, Tel Litwinsky, Israel
- Italy (2):
  - Instituto G. Gaslini, Genova
  - A. Bianchi Bonomi Hemophilia Center, Milan
- Nara Medical University, Nara, Japan
- University Hospital Utrecht, Utrecht, Netherlands
- Malmo University Hospital, Malmo, Sweden
- Changhua Christian Hospital, Chunghua City, Changhua, Taiwan